CLINICAL TRIAL: NCT03420950
Title: Drug Order for Rapid Sequence Intubation in Emergency Department Intubation
Brief Title: Drug Order for Rapid Sequence Intubation
Acronym: DO-RSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Brian Driver, Director of Clinical Research, Dept of Emergency Medicine, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 17-4432
Record Dates: First submitted 2018-01-28; First posted 2018-02-05 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The nurse administering the drug is not blinded, but the outcome assessor and physician performing the intubation are blinded to drug order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedative first (Other): Rapid sequence intubation: sedative first
  Interventions: Other: Rapid sequence intubation: sedative first
- Paralytic agent first (Other): Rapid sequence intubation: paralytic first
  Interventions: Other: Rapid sequence intubation: paralytic first

INTERVENTIONS:
Other: Rapid sequence intubation: sedative first — Sedative first
  Arms: Sedative first
Other: Rapid sequence intubation: paralytic first — Paralytic first
  Arms: Paralytic agent first

SUMMARY:
This is a randomized, blinded trial comparing the order of drug administration for rapid sequence intubation in the Emergency Department.

DETAILED DESCRIPTION:
Based on data (excluding outliers) from protocol 16-4146, the intubation time with the paralytic and sedative first administered is 86 s, and 93 s, respectively, with a standard deviation of approximately 25-30 s. Using these assumptions, 470 patients (235 per group) will need to be enrolled to detect an 7 s absolute difference between groups with 80% power.

Because a greater difference is anticipated in those who receive rocuronium rather than succinylcholine (because succinylcholine takes action faster), goal enrollment is 470 patients who receive rocuronium as the paralytic who are intubated successfully on the first attempt. The total enrollment will be higher, accounting for those who receive succinylcholine and those who are not successful on the first attempt. The data for those who receive succinylcholine first will be reported and is planned to be used to determine the feasibility of a future trial.

The primary group of analysis will be those receiving rocuronium, because this medication acts somewhat slower than succinylcholine. Patients who receive either drug will be analyzed, but it is pre-specified that the group of interest are those receiving rocuronium.

The primary outcome, first intubation attempt duration, and apnea duration will be measured only in those with a successful first attempt because these timing events will be confounded by attempt failure; in these cases the altered duration will have more to do with device or patient characteristics than with drug order.

The remainder of the outcomes will be measured in all enrolled subjects in an intention to treat analysis.

An analysis for patients by RSI drug order actually received, regardless of treatment allocation, will also be presented.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be undergoing orotracheal intubation in the Emergency Department
* The patient must be receiving both a sedative and paralytic immediately prior to intubation (i.e. undergoing rapid sequence intubation).
* The patient must be presumed to be 18 years of age or older at the time of enrollment.

Exclusion Criteria:

* Prisoner or in custody
* Known or suspected to be pregnant, based on the opinion of the attending physician.
* Intubation performed by a physician assistant (this is rarely done in our ED; each physician assistant intubates less than twice per year, so the intubation outcomes would hinge more on their experience rather than drug order).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Time elapsed from drug administration to intubation attempt end | 5 minutes
  The primary outcome will be time from complete administration of the first medication to successful first attempt intubation. This timing period will begin when the first RSI agent is completely administered and end when the laryngoscope blade is removed from the mouth. Attempts that are not successful on the first attempt will be excluded from the primary outcome measure because the time to intubation will be confounded by the failure; in these cases the altered duration will have more to do with device or patient characteristics than with drug order.

SECONDARY OUTCOMES:
Duration of first intubation attempt | 5 minutes
  Defined as the time elapsed between inserting and removing the laryngoscope blade from the mouth. The primary outcome, duration of the first intubation attempt, and apnea duration will only be measured in those with a successful first attempt.
Hypoxemia | 5 minutes
  Oxygen saturation < 90%, during the time interval between the start of the intubation attempt and 1 minute following completion of the attempt.
Best laryngeal view | 5 minutes
  Cormack-Lehane grade
Best laryngeal view | 5 minutes
  Percent of glottic opening
First intubation attempt success | 5 minutes
  Defined as successful intubation with a single insertion of the laryngoscope, regardless of the number of passages of the endotracheal tube or bougie.

OTHER OUTCOMES:
Memory of intubation | 1 week (approximately)
  A structured questionnaire will be administered to patients after extubation. We will attempt to approach all enrolled patients, but realize that some will be unreachable due to death, head injury, rapid discharge from the hospital, and other reason.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Driver, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided